CLINICAL TRIAL: NCT06303713
Title: LuCarbo - a Phase 1a/1b Study of 177Lu-PSMA-617 Plus Carboplatin in Metastatic Castrate-resistant Prostate Cancer
Brief Title: LuCarbo - a Study of 177Lu-PSMA-617 Plus Carboplatin in Metastatic Castrate-resistant Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Praful Ravi, MB BCHir, MRCP, Sponsor Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23-693
Record Dates: First submitted 2024-02-27; First posted 2024-03-12 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer; Metastatic Prostate Cancer; Metastatic Castration-resistant Prostate Cancer
Keywords: Prostate Cancer; Metastatic Prostate Cancer; Metastatic Castration-resistant Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Carboplatin; Platinum; Pluvicto

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1A: Dose Escalation (Experimental): Participants will be enrolled in a 3+3 dose escalation design to establish a maximum tolerated dose (MTD) of carboplatin, starting at Dose Level 1 and escalating to Dose Level 2 or 3.
  * Baseline visit.
  * Day 1 of Cycles 3 and 5: Tumor assessment radiologic scans.
  * Cycle 1 through End of Treatment:
    * Days 1 and 22 of 42-day cycle: Predetermined dose of carboplatin every 3 weeks for a maximum of up to 6 cycles.
    * Day 2 of 42-day cycle: Predetermined dose of 177Lu-PSMA-617 every 6 weeks for a maximum of up to 6 cycles.
  * End of treatment visit.
  * Follow up visits in-office or via telephone. If 0 out of 3 participants experience a dose-limiting toxicity (DLT), the study will proceed to the next dose level. If 1 or more participants experience a DLT, this dose level is declared the MTD and study will not proceed to expansion. If 1 out of 6 participants at the highest dose level experience DLTs, this is the recommended Phase 1B dose.
  Interventions: Drug: Carboplatin; Drug: 177Lu-PSMA-617
- Phase 1B: Dose Expansion (Experimental): 19 additional participants will be enrolled at the RP2D of carboplatin and will complete:
  * Baseline visit.
  * Day 1 of Cycles 3 and 5: Tumor assessment radiologic scans.
  * Tumor biopsy at baseline and at 12 weeks.
  * Cycle 1 through End of Treatment:
    * Days 1 and 22 of 42 day cycle: Predetermined dose of carboplatin every 3 weeks for a maximum of up to 6 cycles.
    * Day 2 of 42 day cycle: Predetermined dose of 177Lu-PSMA-617 every 6 weeks for a maximum of up to 6 cycles.
  * End of treatment visit.
  * Follow up visits in-office or via telephone.
  Interventions: Drug: Carboplatin; Drug: 177Lu-PSMA-617

INTERVENTIONS:
Drug: Carboplatin — Platinum coordination compound, premixed aqueous solution of 10mg/ML, via intravenous (into the vein) infusion per protocol.
  Other Names: C6H12N2O4Pt; Platinum, diammine [1,1-cyclobutanedicarboxylato(2-)- O,O']-, (SP-4-2)
Drug: 177Lu-PSMA-617 — Radioligand therapy, single-dose vial, via intravenous (into the vein) infusion per protocol.
  Other Names: Pluvicto; Lutetium Lu 177 vipivotide tetraxetan; C49H71N9O16

SUMMARY:
The purpose of this study is to see whether the combination of a chemotherapy drug, carboplatin, along with the radioligand treatment, 177Lu-PSMA-617, is safe in treating prostate cancer and whether the combination is effective in shrinking or preventing growth of prostate cancer.

The names of the study drugs used in this research study are:

* Carboplatin (A type of chemotherapy)
* 177Lu-PSMA-617 (A type of radioligand therapy)

DETAILED DESCRIPTION:
This is a phase 1 dose-escalation and dose-expansion trial of carboplatin in combination with 177Lu-PSMA-617 in participants with metastatic castrate-resistant prostate cancer (mCRPC). The study will take place in two parts: Phase 1a to define the recommended phase 2 dose (RP2D) and Phase 1b to further assess safety and preliminary clinical activity of the combination regimen.

The U.S. Food and Drug Administration (FDA) has not approved carboplatin for prostate cancer but it has been approved for other uses.

The U.S. FDA has approved 177Lu-PSMA-617 as a treatment option for prostate cancer.

The research study procedures include screening for eligibility and study treatment visits, tumor biopsies, x-rays, Computerized Tomography (CT) scans, Magnetic Resonance Imaging (MRI) scans, Positron Emission Tomography (PET) scans, and blood tests.

It is expected that about 35 people will take part in this research study.

Novartis is supporting this research study by providing 177Lu-PSMA-617, as well as research funding.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed prostate adenocarcinoma without histologic variants comprising >50% of the sample as determined by pathology review at an academic medical center; men without histologic or cytologic confirmation are eligible provided there is unequivocal evidence of prostate cancer (eg. very high PSA) in the view of the treating physician.
* Age ≥ 18years. Children under age 18 are excluded as prostate cancer is a disease of adults.
* Progressive disease at study entry, as defined by either one of the following:

  * Sequence of at least 2 rising PSA values at a minimum of 1-week intervals with the last result being ≥1.0 ng/mL if confirmed PSA rise is the only indication of progression. Patients who received an anti-androgen (flutamide, bicalutamide or nilutamide) must have PSA progression ≥4 weeks after the last dose.
  * Radiographic progression per RECIST 1.1 for soft tissue and/or per PCWG3 for bone (i.e. appearance of ≥2 new bone lesions), with or without PSA progression.
* Presence of ≥1 metastatic lesion metastatic lesion present on baseline CT, MRI, or bone scan imaging obtained ≤28 days prior to beginning study therapy.
* Prior receipt of at least one taxane chemotherapy (docetaxel or cabazitaxel) and at least one ARPI (abiraterone, enzalutamide, apalutamide or darolutamide) in the localized, recurrent or metastatic setting. Prior treatment with a PARP inhibitor(s) is permitted. Prior treatment with Ra-223 is permitted, providing that the last dose of Ra-223 was ≥90 days prior to study entry.
* Presence of ≥1 PSMA-avid lesion (with uptake > liver) on baseline/screening 68GaPSMA-11 PSMA-PET.
* Serum testosterone level must be ≤50ng/dL (1.73 nmol/L) at the screening visit. Participants who have not undergone bilateral orchiectomy are required to continue LHRH/GnRH agonists/antagonists) throughout the study. Use of relugolix is permitted.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A).
* Adequate organ and marrow function as per the below table:

  --System Laboratory Value
* Hematologic

  * ANC ≥1.5×109/L
  * Platelets ≥100×109/L
  * Hemoglobin ≥9g/dL (≥90g/L), independent of transfusions
* Hepatic

  * Total bilirubin ≤1.5 × ULN OR <2 × ULN if known or suspected Gilbert's syndrome
  * ALT and AST ≤3 × ULN OR ≤5 × ULN if liver metastases present
* Renal

  --eGFR ≥30 mL/min/1.73 m2 (based on Cockcroft-Gault formula OR 24 hour urine collection
* Presence of a recurrent/metastatic lesion (bone or soft tissue) amenable to image-guided percutaneous biopsy adequate for next generation sequencing (NGS), and planned to undergo core biopsy after trial registration but prior to cycle 1 day 1 of therapy.

Confirmation of adequacy of this biopsy material for NGS is NOT required for initiation of therapy.

* Willingness to undergo core biopsy of a recurrent/metastatic lesion adequate for NGS after approximately 12 weeks of study treatment.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* The effects of 177Lu-PSMA-617 and carboplatin on the developing human fetus are unknown. For this reason and because chemotherapies and radioligand therapies are known to be teratogenic, men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Men treated or enrolled on this protocol must also agree to use adequate contraception for the duration of study participation, and at least 14 weeks following the last dose of 177Lu-PSMA-617.Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform her treating physician immediately. Female partners of child-bearing potential should also use highly effective birth control methods throughout the male participant's study treatment and for at least 14 weeks following the last dose of 177Lu-PSMA-617.
* Ability to understand and the willingness to sign a written informed consent document. (Providing consents in as many languages as possible is encouraged)

Exclusion Criteria

* Participants who have had chemotherapy or radiotherapy within 4 weeks prior to planned cycle 1 day 1 of study treatment.
* Participants who have received anti-neoplastic intervention or experimental antineoplastic therapy within 14 days of planned cycle 1 day 1 of study therapy.
* Participants who are receiving any other investigational agents.
* Participants who have previously received 177Lu-PSMA-617.
* Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 177Lu-PSMA-617 and carboplatin.
* Participants with untreated brain metastases. Participants with treated brain metastases are eligible if follow-up brain imaging at least 4 weeks after central nervous system (CNS)-directed therapy shows no evidence of progression and ongoing corticosteroids are not required. Participants with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy.
* Symptomatic cord compression, or clinical or radiologic findings indicative of impending cord compression.
* Concurrent active malignancy whose natural history or treatment has the potential to interfere with safety or efficacy assessment of the investigational regimen. Patients with non-melanomatous skin cancer, superficial bladder cancer, cancer not needing active therapy for at least 2 years, cancer for which the treating investigator deems the subject to be in remission, or any prior malignancy that was treated with curative intent (no evidence of disease for at least 3 years) are permitted to enroll.
* The participant has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 37 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2026-07-19 (Estimated); Study Completion 2026-07-19 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) or the Recommended Phase 2 dose (RP2D) of carboplatin administered in combination with 177Lu-PSMA-617 | First 6 weeks of treatment
  The RP2D will be the highest administered dose level with ≤1 dose-limiting toxicities (DLTs) out of 6 treated patients.

SECONDARY OUTCOMES:
PSA response rate (PSA reduction by ≥50% from baseline). | Through study completion, an average of 1 year
  PSA response rate is defined as the proportion of participants achieving ≥50% reduction in PSA from baseline during study treatment
Overall Response Rate (ORR) | Through study completion, an average of 1 year
  The overall response rate (ORR) is defined as the proportion of participants achieving either PSA reduction by ≥50 or complete response (CR) or partial response (PR) based on RECISTv1.1 criteria.
Radiographic Progression-Free Survival (rPFS) | Through study completion, an average of 1 year
  rPFS is defined as the time from the start of the treatment to the earlier of progression or death due to any cause. Progression is defined per RECIST 1.1 for soft tissue and PCWG3 for bone lesions. Participants alive without disease progression are censored at date of last disease evaluation.
Overall Survival (OS) | Through study completion, an average of 1 year
  Overall Survival (OS) based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.

CONTACTS AND LOCATIONS:
Overall Officials: Praful Ravi, MB BCHir, MRCP, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu.